CLINICAL TRIAL: NCT01422928
Title: Does Radiation Therapy Adversely Affect the Immune System, and Can Acupuncture Ameliorate the Effect? A Pilot Study
Brief Title: Acupuncture for the Immune System in Radiation Cancer Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was not approved by research ethics board.
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: BC Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCCA- H10-02105
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Gastrointestinal Neoplasms; Urogenital Neoplasms
Keywords: Radiotherapy; Acupuncture; Immune System
MeSH Terms: conditions — Gastrointestinal Neoplasms; Urogenital Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment (No Intervention): Patients receiving standard radiation therapy for gastrointestinal or urogenital cancers.
  All subjects will be asked to give 20 mL of blood and complete the Edmonton Symptom Assessment Form (ESAS) on 3 occasions:
  * before radiation
  * at 1st follow up 4-10 weeks after radiation completion
  * at second follow up 6 months after 1st follow up
- Acupuncture (Experimental): Patients receiving standard radiation therapy for gastrointestinal or urogenital cancers with concurrent acupuncture once a week for 4 weeks.
  All subjects will be asked to give 20 mL of blood and complete the Edmonton Symptom Assessment Form (ESAS) on 3 occasions:
  * before radiation
  * at 1st follow up 4-10 weeks after radiation completion
  * at second follow up 6 months after 1st follow up
  Interventions: Procedure: Medical Acupuncture

INTERVENTIONS:
Procedure: Medical Acupuncture — Subjects will be asked to report symptom concerns. Subjects are requested to wear loose clothing as most acupoints lie at or distal to the elbow and knee.
  Sterile single use steel needles (ITO Adiquip 0.25 x 4.0 cm) will be inserted to a depth of 1 - 2 cm at acupoints thought to impact positively on the immune system. An ITO ES-160 Electrostimulator will be used to mimic the "pecking" technique of manual stimulation. Following needle insertion by the acupuncturist, a nurse or acupuncture student may assist by attaching electrodes to provide electrical stimulation. A 0.3 ms duration, 4 HZ, alternating current will be delivered with voltage set just below the pain threshold of the patient. After 20 minutes, the needles will be removed. Acupoints will include:
  * GV.14
  * LI.11 (bilateral)
  * SP.6 (bilateral)
  * SP.10 (bilateral)
  * ST.36 (bilateral)
  Additional points may be added based on the symptom concerns reported.
  Arms: Acupuncture

SUMMARY:
Purpose/Goal: To investigate how long course radiation therapy (RT), both with or without chemotherapy, affects the immune system, and to determine if acupuncture can modify these effects in patients undergoing curative radiation therapy for gastrointestinal (GI) or genitourinary (GU) cancers.

Clinical or Research Questions:

1. Does RT reduce immune biomarkers in treated subjects?
2. Which biomarkers are most affected by treatment?
3. Is acupuncture a feasible option to help ameliorate any biomarker effects?
4. Does RT affect subject symptoms?
5. Is acupuncture a feasible option to help ameliorate any symptom effects?

DETAILED DESCRIPTION:
Research indicates that patients undergoing curative RT for various cancers experience adverse immune effects, as indicated by reduced biomarker levels and activity. RT has been observed to cause a striking reduction in total lymphocyte count, affecting mainly the T-cells. Furthermore, the reduction in the lymphocyte count after RT has been correlated with poorer outcome for bladder cancer, head and neck cancer, uterine cancer, and brain metastases.

Research into the use of complementary and alternative medicine (CAM) has been conducted to determine the utility of these treatments in addressing the unmet needs of many patients with cancer. There is preliminary evidence that acupuncture, in particular, is successful at improving many cancer and treatment associated effects. Earlier studies have indicated that acupuncture can play a role in regulating immune system response to various morbidities, including chemotherapy induced immunosuppression. However, little research has examined is potential for radiation therapy patients

This pilot study aims to assess a wide range of general immune biomarkers to identify biomarkers most affected by RT. Through use of a symptom assessment survey, changes in self reported symptoms will also be recorded. The feasibility of acupuncture as a strategy to ameliorate any adverse immune or symptom effects will also be examined. This information could be very useful in planning future studies on RT and the immune system, or the potential immune benefits of acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* patients who will receive ≥ 4 weeks of curative intent long course RT for a GI or GU malignancy
* patients may or may not have received / be receiving adjuvant chemotherapy
* anticipated survival of at least 12 months
* able to visit the BCCA VIC for treatment and 2 follow up visits

Exclusion Criteria:

* scheduled to receive RT for a period of less than 4 weeks
* expected survival period is less than 12 months
* are on anticoagulants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Changes in immune biomarker levels | As measured using 3 blood samples collected: before radiation; at 1st follow up 4-10 weeks after radiation completion; at second follow up 6 months after 1st follow up
  Change in 21 immune cell types after RT (levels before RT - levels 1st follow up) will be analyzed for controls (to determine if RT reduces immune markers) and experimentals (to determine if acupuncture ameliorates RT effects). Results will be analyzed to determine which biomarkers experienced the largest changes for controls (to identify biomarkers affected by RT) and experimentals (to determine which biomarkers are particularly improved by acupuncture). Change in cell levels during follow up (levels 1st follow up - levels 2nd follow up), will be analyzed to determine duration of changes.

SECONDARY OUTCOMES:
Changes in Symptom Scores | As measured using the Edmonton Symptom Assessment Scores (ESAS) completed: before radiation; at 1st follow up 4-10 weeks after radiation completion; at second follow up 6 months after 1st follow up
  The change in ESAS following treatment (ESAS before treatment - ESAS at first follow up) will be analyzed for control subjects (to determine if RT affects subject symptoms) and experimental subjects (to determine if acupuncture ameliorates any symptom effects). For each subject, results will be analyzed for the change in the total ESAS after treatment, as well as the largest change in ESAS for any single symptom. Also, change in ESAS in the follow up period (ESAS at first follow up - ESAS at second follow up), will be analyzed in order to determine the duration of any changes.

CONTACTS AND LOCATIONS:
Overall Officials: Jan T W Lim, MD, Principal Investigator — BC Cancer Agency and University of British Columbia
Locations (1):
- BC Cancer Agency - Vancouver Island Centre, Victoria, British Columbia, Canada